CLINICAL TRIAL: NCT01435616
Title: A Comparison of LY2605541 Versus Insulin Glargine as Basal Insulin Treatment in Combination With Oral Anti-Hyperglycemia Medications in Insulin-Naive Patients With Type 2 Diabetes Mellitus: A Double-Blind, Randomized Study
Brief Title: A Study in Patients With Type 2 Diabetes Mellitus
Acronym: IMAGINE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12141; I2R-MC-BIAJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-09-09; First posted 2011-09-16 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes mellitus; type 2 diabetes mellitus; insulin naive; insulin treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Insulin Glargine; LY2605541

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LY2605541 (Experimental): LY2605541 titrated based on blood glucose readings, administered subcutaneously (SC), once daily in combination with at least 2 pre-study oral antihyperglycemic medications (OAMs) prescribed by the personal physician, for 52 or 78 weeks
  Interventions: Drug: LY2605541
- Glargine (Active Comparator): Glargine titrated based on blood glucose readings, administered SC, once daily in combination with at least 2 pre-study OAMs prescribed by the personal physician, for 52 or 78 weeks
  Interventions: Drug: Glargine

INTERVENTIONS:
Drug: Glargine
  Arms: Glargine
Drug: LY2605541
  Arms: LY2605541

SUMMARY:
The purpose of this study is:

* To compare blood sugar control on LY2605541 with insulin glargine after 52 weeks of treatment.
* To compare the rate of night time low blood sugar episodes on LY2605541 with insulin glargine during 52 weeks of treatment.
* To compare the number of participants on LY2605541 reaching blood sugar targets without low blood sugar episodes at night to those taking insulin glargine after 52 weeks of treatment.
* To compare the rate of low blood sugar episodes on LY2605541 with insulin glargine after 52 weeks of treatment

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes mellitus, not treated with insulin, for at least 1 year prior to the study
* Have been receiving at least 2 OAMs for at least 3 months before entering the study
* Have a hemoglobin A1c (HbA1c) value between 7.0% and 11.0%, inclusive, at screening
* Are capable of and willing to inject insulin with a vial and syringe and perform self blood glucose monitoring
* Women of childbearing potential only: are not breastfeeding, have a negative pregnancy test at the time of screening and randomization, intend to not become pregnant during the trial, have practiced a reliable method of birth control for at least 6 weeks prior to screening, and agree to use a reliable method of birth control during the study and until 2 weeks following the last dose of study drug

Exclusion Criteria:

* Have used insulin therapy (outside of pregnancy) anytime in the past 2 years, except for short-term treatment of acute conditions, and up to a maximum of 4 continuous weeks
* Use of rosiglitazone, pramlintide, or glucagon-like peptide 1 (GLP-1) receptor agonist (for example, exenatide, exenatide once weekly, or liraglutide) concurrently or within 3 months prior to screening
* Are currently taking, or have taken within the 3 months preceding screening, medications to promote weight loss
* Have had any episodes of severe hypoglycemia within 6 months prior to screening
* Have had 1 or more episodes of ketoacidosis or hyperosmolar state/coma in the 6 months prior to the study
* Have cardiac disease with functional status that is New York Heart Association Class III or IV (per New York Heart Association [NYHA] Cardiac Disease Classification)
* Have a history of renal transplantation, or are currently receiving renal dialysis or have serum creatinine greater or equal than 2 milligrams per deciliter (mg/dL)
* Have obvious clinical signs or symptoms of liver disease (excluding non- alcoholic fatty liver disease [NAFLD]), acute or chronic hepatitis, non-alcoholic steatohepatitis (NASH), or elevated liver enzyme measurements at screening
* Have had a blood transfusion or severe blood loss within 3 months prior to screening or have known hemoglobinopathy, hemolytic anemia or sickle cell anemia, or any other traits of hemoglobin abnormalities known to interfere with the measurement of HbA1c
* Have active or untreated malignancy or have been in remission from clinically significant malignancy for less than 5 years
* Have fasting or non-fasting triglycerides greater than 400 mg/dL (greater than 4.5 millimoles per liter [mmol/L]) at screening
* Are using lipid-lowering medication at a dose that has not been stable for 90 days prior to screening
* Are using niacin preparations as a lipid lowering medication and bile acid sequestrants within 90 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1538 (Actual)
Dates: Start 2011-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (167):
- United States (66):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anniston, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mobile, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chandler, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesa, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tempe, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenbrae, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntington Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mission Viejo, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Northridge, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Springs, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Mateo, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tustin, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winter Haven, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Decatur, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Meridian, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangor, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haverhill, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gallipolis, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Perrysburg, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Corvallis, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beaver, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Downingtown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lansdale, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Levittown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pottstown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greer, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Myrtle Beach, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bristol, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Hill, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marshall, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sugar Land, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bountiful, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clinton, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ogden, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olympia, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Port Orchard, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
- Argentina (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mar del Plata
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Merewether, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Keswick, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Box Hill, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fremantle, Western Australia
- Brazil (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marília
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Setor Oeste/Goiania
- Canada (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Victoria, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Etobicoke, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Markham, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Laval, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pointe-Claire, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
- Finland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oulu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seinäjoki
- Germany (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dippoldiswalde
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Friedrichsthal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Furth im Wald
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ludwigshafen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saarbrücken
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Schweinfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sulzbach
- Greece (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ampelokipoi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Hungary (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Makó
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salgótarján
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sopron
- Israel (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beersheba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raanana
- Italy (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carpi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Castellanza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Foggia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Forlì
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sesto San Giovanni
- Lithuania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Utena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vilnius
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coatzacoalcos
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Auckland, New Zealand
- Poland (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kamieniec Ząbkowicki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Katowice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ruda Śląska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tychy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Puerto Rico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hato Rey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
- Romania (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oradea
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ploieşti
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reşiţa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
- Russia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cheboksary
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kazan'
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kursk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Novosibirsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- Slovakia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Šaľa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vranov nad Topľou
- South Africa (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paarl
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Somerset West
- Spain (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pozuelo de Alarcón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Requena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toledo
- Turkey (Türkiye) (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gaziantep
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hatay
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Izmir
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kayseri
- United Kingdom (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mortimer, Berks
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leicester, Leicestershire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guildford, Surrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Swansea, Wales

REFERENCES:
- [Derived] Qu Y, White RD, Ruberg SJ. Accurate Collection of Reasons for Treatment Discontinuation to Better Define Estimands in Clinical Trials. Ther Innov Regul Sci. 2023 May;57(3):521-528. doi: 10.1007/s43441-022-00491-0. Epub 2022 Dec 21. PMID 36542287
- [Derived] Sanyal A, Cusi K, Hartman ML, Zhang S, Bastyr EJ 3rd, Bue-Valleskey JM, Chang AM, Haupt A, Jacober SJ, Konrad RJ, Zhang Q, Hoogwerf BJ. Cytokeratin-18 and enhanced liver fibrosis scores in type 1 and type 2 diabetes and effects of two different insulins. J Investig Med. 2018 Mar;66(3):661-668. doi: 10.1136/jim-2017-000609. Epub 2017 Nov 21. PMID 29167192
- [Derived] Orchard TJ, Cariou B, Connelly MA, Otvos JD, Zhang S, Antalis CJ, Ivanyi T, Hoogwerf BJ. The effects of basal insulin peglispro vs. insulin glargine on lipoprotein particles by NMR and liver fat content by MRI in patients with diabetes. Cardiovasc Diabetol. 2017 Jun 6;16(1):73. doi: 10.1186/s12933-017-0555-1. PMID 28587667
- [Derived] Cusi K, Sanyal AJ, Zhang S, Hartman ML, Bue-Valleskey JM, Hoogwerf BJ, Haupt A. Non-alcoholic fatty liver disease (NAFLD) prevalence and its metabolic associations in patients with type 1 diabetes and type 2 diabetes. Diabetes Obes Metab. 2017 Nov;19(11):1630-1634. doi: 10.1111/dom.12973. Epub 2017 Jun 22. PMID 28417532

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LY2605541 | Glargine
Started | 1003 | 535
Received at Least 1 Dose of Study Drug | 1003 | 535
Completed | 832 | 455
Not Completed | 171 | 80
Not completed — Adverse Event | 39 | 21
Not completed — Death | 7 | 2
Not completed — Lost to Follow-up | 22 | 13
Not completed — Protocol Violation | 16 | 13
Not completed — Withdrawal by Subject | 66 | 24
Not completed — Physician Decision | 20 | 7
Not completed — Sponsor Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- LY2605541: LY2605541 titrated based on blood glucose readings, administered SC, once daily in combination with at least 2 pre-study OAMs prescribed by the personal physician, for 52 or 78 weeks
- Total: Total of all reporting groups
Arm/Group | LY2605541 | Glargine | Total
Number analyzed (Participants) | 1003 | 535 | 1538
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.80 (9.85) | 59.35 (9.80) | 58.99 (9.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 453 | 227 | 680
  Male | 550 | 308 | 858
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 201 | 96 | 297
  Not Hispanic or Latino | 648 | 355 | 1003
  Unknown or Not Reported | 154 | 84 | 238
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 24 | 15 | 39
  Asian | 25 | 12 | 37
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Black or African American | 68 | 34 | 102
  White | 875 | 469 | 1344
  More than one race | 8 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 371 | 188 | 559
  Slovakia | 12 | 10 | 22
  Greece | 18 | 12 | 30
  Finland | 6 | 7 | 13
  Spain | 35 | 18 | 53
  Turkey | 7 | 4 | 11
  Lithuania | 8 | 4 | 12
  Israel | 16 | 8 | 24
  Russia | 32 | 18 | 50
  Italy | 24 | 13 | 37
  United Kingdom | 12 | 5 | 17
  Hungary | 69 | 33 | 102
  Mexico | 24 | 16 | 40
  Puerto Rico | 39 | 19 | 58
  Canada | 16 | 11 | 27
  Argentina | 67 | 34 | 101
  Brazil | 20 | 10 | 30
  Poland | 67 | 32 | 99
  Romania | 40 | 22 | 62
  Australia | 27 | 18 | 45
  South Africa | 11 | 4 | 15
  Germany | 63 | 36 | 99
  New Zealand | 10 | 9 | 19
  Czechia | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 52 Week Endpoint in Hemoglobin A1c (HbA1c)
Description: HbA1C is a test that measures a person's average blood glucose level over the past 2 to 3 months. Least Squares (LS) means were calculated using a mixed model repeated measures (MMRM) with baseline HbA1c measurement, stratification factors (country, low density lipoprotein-cholesterol [LDL-C, < 100 milligrams per deciliter {mg/dL} and ≥ 100 mg/dL] and sulfonylurea [SU]/meglitinide use), visit, treatment, and visit-by-treatment interaction as fixed effects.
Time Frame: Baseline, 52 weeks
Population: All participants who were randomized, had at least 1 dose of study medication, and at least 1 post-baseline HbA1c measurement.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Groups:
- LY2605541: LY2605541 titrated based on blood glucose readings, administered SC, once daily in combination with at least 2 pre-study OAMs prescribed by the personal physician, for 52 weeks
- Glargine: Glargine titrated based on blood glucose readings, administered SC, once daily in combination with at least 2 pre-study OAMs prescribed by the personal physician, for 52 weeks
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 989 | 523
percentage of HbA1c | -1.55 (0.03) | -1.25 (0.04)

2. Secondary Outcome: Rate of Total and Nocturnal Hypoglycemia Events
Description: Hypoglycemia is a condition that occurs when a person's blood glucose level is lower than the normal range (less than or equal to 70 milligrams per deciliter [mg/dL] or less than 3.9 millimoles per liter [mmol/L]). Total hypoglycemia refers to an event that meets the criteria for documented symptomatic hypoglycemia, asymptomatic hypoglycemia, probable symptomatic hypoglycemia, unspecified hypoglycemia, or severe hypoglycemia. Nocturnal hypoglycemia refers to any total hypoglycemic event that occurs between bedtime and waking. Group mean (listed as LS means below) rates of total and nocturnal hypoglycemia were calculated using a negative binomial regression model (number of episodes = treatment + SU/meglitinide use + baseline hypoglycemia event rate, with log [exposure per 30 days] as the offset variable in the model).
Time Frame: Baseline to 52 weeks
Population: All participants who were randomized, who received at least 1 dose of study drug, and had evaluable total and/or nocturnal event data.
Measure: Least Squares Mean (Standard Error); unit: episodes/participant/30 days
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 1001 | 535
episodes/participant/30 days
  Rate of total hypoglycemia events | 1.16 (0.06) | 1.21 (0.07)
  Rate of nocturnal hypoglycemia events | 0.30 (0.02) | 0.40 (0.03)

3. Secondary Outcome: Percentage of Participants With Hemoglobin A1c Equal or Less Than 6.5% and Less Than 7.0 %
Description: The percentage of participants was calculated by dividing the number of participants reaching target HbA1c by the total number of participants analyzed, multiplied by 100.
Time Frame: 52 weeks
Population: All participants who were randomized, received at least 1 dose of study drug, and had at least 1 post-baseline HbA1c measurement.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 989 | 523
percentage of participants
  HbA1c ≤ 6.5% | 36.1 | 23.9
  HbA1c < 7.0% | 57.6 | 42.8

4. Secondary Outcome: Fasting Serum Glucose (By Laboratory Measurement)
Description: LS means were calculated using a MMRM with baseline fasting serum glucose measurement, stratification factors (country, HbA1c, LDL-C [< 100 mg/dL and ≥ 100 mg/dL], and SU/meglitinide use), treatment, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: 52 weeks
Population: All participants who were randomized, received at least 1 dose of study drug, and had evaluable fasting serum glucose data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 986 | 521
mg/dL | 114.93 (1.24) | 120.13 (1.70)

5. Secondary Outcome: Fasting Blood Glucose (By Participant Self-monitored Blood Glucose Readings)
Description: LS means were calculated using a MMRM with baseline fasting blood glucose measurement, stratification factors (country, HbA1c, LDL-C [< 100 mg/dL and ≥ 100 mg/dL], and SU/meglitinide use), treatment, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: 52 weeks
Population: All participants who were randomized, received at least 1 dose of study drug, and had evaluable fasting blood glucose data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 994 | 528
mg/dL | 112.57 (0.82) | 112.00 (1.12)

6. Secondary Outcome: 6 Point Self-monitored Blood Glucose (SMBG)
Description: Six-point SMBG profiles were obtained at pre-morning meal (fasting), pre-midday meal (lunch), pre-evening meal (dinner), bedtime, approximately 0300 hours, and pre-morning meal (fasting) the next day. Six-point SMBG profiles were obtained over 2 nonconsecutive days within the week prior to the next office visit. LS means were calculated using a MMRM with baseline blood glucose measurement, stratification factors (country, HbA1c, LDL-C [< 100 mg/dL and ≥ 100 mg/dL], and SU/meglitinide use), treatment, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: 52 weeks
Population: All participants who were randomized, received at least 1 dose of study drug, and had evaluable SMBG data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 943 | 499
mg/dL
  Pre-morning meal | 112.81 (0.96) | 112.26 (1.31)
  Pre-midday meal: number analyzed (Participants) | 925 | 494
  Pre-midday meal | 127.65 (1.36) | 134.52 (1.86)
  Pre-evening meal: number analyzed (Participants) | 928 | 494
  Pre-evening meal | 133.94 (1.40) | 142.58 (1.91)
  Bedtime: number analyzed (Participants) | 911 | 486
  Bedtime | 151.37 (1.54) | 155.19 (2.10)
  0300 hours: number analyzed (Participants) | 909 | 466
  0300 hours | 120.35 (1.21) | 118.37 (1.67)
  Pre-morning meal (next day): number analyzed (Participants) | 939 | 494
  Pre-morning meal (next day) | 111.11 (0.89) | 109.19 (1.23)

7. Secondary Outcome: Change From Baseline to 52 Weeks in Body Weight
Description: LS means were calculated using a MMRM with baseline body weight measurement, stratification factors (country, HbA1c, LDL-C [< 100 mg/dL and ≥ 100 mg/dL], and SU/meglitinide use), treatment, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, 52 weeks
Population: All participants who were randomized, who received at least 1 dose of study drug, and had evaluable body weight data.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 985 | 522
kilograms (kg) | 2.06 (0.15) | 2.57 (0.21)

8. Secondary Outcome: Hemoglobin A1c
Description: HbA1c is a test that measures a person's average blood glucose level over the past 2 to 3 months. LS means were calculated using a MMRM with baseline HbA1C measurement, stratification factors (country, HbA1c, LDL-C [< 100 mg/dL and ≥ 100 mg/dL], and SU/meglitinide use), treatment, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: 52 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 989 | 523
percentage of HbA1c | 6.91 (0.03) | 7.21 (0.04)

9. Secondary Outcome: Insulin Dose Per Body Weight
Description: LS means were calculated using a MMRM with baseline insulin dose measurement, stratification factors (country, HbA1c, LDL-C [< 100 mg/dL and ≥ 100 mg/dL], and SU/meglitinide use), treatment, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: 52 weeks
Population: All participants who were randomized, received at least 1 dose of study drug, and had evaluable insulin dose data.
Measure: Least Squares Mean (Standard Error); unit: units of insulin/kg body weight
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 1001 | 532
units of insulin/kg body weight | 0.45 (0.01) | 0.42 (0.01)

10. Secondary Outcome: Number of Insulin Dose Adjustments to Steady-State
Description: Insulin doses were adjusted according to an algorithm (adapted from Riddle et al. 2003) during the first 26 weeks of the study and thereafter according to investigator judgment. Steady-state was defined as the first local maximum dose (maximum of moving 4-week interval) of LY2605541 or glargine within the window of +/- 2 weeks. The number of dose adjustments to steady-state was the total number of dose changes until steady-state was reached. LS means were calculated using a MMRM with baseline insulin dose measurement, stratification factors (country, HbA1c, LDL-C [< 100 mg/dL and ≥ 100 mg/dL], and SU/meglitinide use), treatment, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline to 52 weeks
Population: All participants who were randomized, received at least 1 dose of study drug, and had evaluable post-baseline insulin data.
Measure: Least Squares Mean (Standard Error); unit: number of insulin dose adjustments
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 1002 | 532
number of insulin dose adjustments | 5.83 (0.12) | 5.25 (0.16)

11. Secondary Outcome: European Quality of Life-5 Dimension (EQ-5D)
Description: The EQ-5D is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows participants to rate their health state in 5 health domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) using a 3-level scale of 1 to 3 (no problem, some problems, and extreme problems). These combinations of attributes are converted into a weighted health-state Index Score according to the United States population-based algorithm. Scores range from -0.11 to 1.0, where a score of 1.0 indicates perfect health. LS means were calculated using a MMRM with baseline stratification factors (country, HbA1c, and SU/meglitinide use), treatment, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: 52 weeks
Population: All participants who were randomized, received at least 1 dose of study drug, and had evaluable EQ-5D data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 892 | 474
units on a scale | 0.88 (0.00) | 0.88 (0.01)

12. Secondary Outcome: Insulin Treatment Satisfaction Questionnaire
Description: The Insulin Treatment Satisfaction Questionnaire (ITSQ) is a validated instrument containing 22 items that assess treatment satisfaction for participants with diabetes who are receiving insulin. The questionnaire measures satisfaction from the following 5 domains: inconvenience of regimen, lifestyle flexibility, glycemic control, hypoglycemic control, and insulin delivery device. Data presented are the transformed total score on a scale of 0 to 100, where higher scores indicate better treatment satisfaction. LS means were calculated using a MMRM with stratification factors (country, HbA1c, and SU/meglitinide use), treatment, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: Up to 52 weeks
Population: All participants who were randomized, received at least 1 dose of study drug, and had evaluable ITSQ data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 966 | 515
units on a scale | 84.73 (0.44) | 85.04 (0.60)

13. Secondary Outcome: Adult Low Blood Sugar Survey
Description: The adult Low Blood Sugar Survey (LBSS) is a validated, participant-reported 33-item questionnaire with items rated on a 5-point Likert scale, where 0 = never and 4 = always. The LBSS measures behaviors to avoid hypoglycemia and its negative consequences (15 items) and worries about hypoglycemia and its negative consequences (18 items). Total score is the sum of all items (range of 0 to 132). Higher total scores reflect greater fear of hypoglycemia. LS means were calculated using an analysis of covariance model (ANCOVA) with baseline LBSS score, stratification factors (country, HbA1c, and SU/meglitinide use), and treatment as fixed effects.
Time Frame: Up to 52 weeks
Population: All participants who were randomized, received at least 1 dose of study drug, and had evaluable LBSS data. Missing endpoints were imputed with the last observation carried forward (LOCF) method, using only post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 899 | 478
units on a scale | 15.09 (0.49) | 14.59 (0.67)

14. Secondary Outcome: Change From Baseline to 52 Weeks in Triglycerides, Low Density Lipoprotein Cholesterol (LDL-C), and High Density Lipoprotein Cholesterol (HDL-C)
Description: LS means were calculated using a MMRM with baseline lipid measurement, stratification factors (country, HbA1c, LDL-C [< 100 mg/dL and ≥ 100 mg/dL], and SU/meglitinide use), treatment, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, 52 weeks
Population: All participants who were randomized, received at least 1 dose of study drug, and had at least 1 post-baseline lipid measurement.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 992 | 528
milligrams per deciliter (mg/dL)
  Triglycerides | 10.60 (2.46) | -7.33 (3.38)
  LDL-C: number analyzed (Participants) | 992 | 527
  LDL-C | 1.44 (0.83) | 1.76 (1.14)
  HDL-C | -1.91 (0.21) | -1.82 (0.29)

15. Secondary Outcome: Percentage of Participants With Equal or Above 2-, and 3-fold Upper Limits of Normal (ULN) for Total Bilirubin
Time Frame: Up to 52 weeks
Population: All participants who were randomized, had at least 1 dose of study drug, and had at least 1 post-baseline total bilirubin measurement.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 994 | 529
percentage of participants
  ≥2-fold ULN | 0.2 | 0.0
  ≥3-fold ULN | 0.1 | 0.0

16. Secondary Outcome: Overall Treatment-Emergent Anti-LY2065541 Antibody Response (TEAR)
Description: The percentage of participants with a TEAR is summarized. TEAR is defined as a change in the anti-LY2605541 antibody level from undetectable at baseline to detectable at baseline, or, for those participants with detectable antibodies at baseline, change to a value with at least a 130% relative increase from baseline. Overall TEAR is defined as one or more TEAR during the specified period.
Time Frame: Baseline to 78 weeks
Population: All participants who were randomized, received at least 1 dose of study drug, and had evaluable TEAR data.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 988 | 521
percentage of participants | 43.0 | 37.8

17. Secondary Outcome: Intra-participant Variability of the Fasting Blood Glucose (FBG)
Description: Intra-participant variability of FBG, which was measured by SMBG, was assessed by the standard deviation of the FBG measurement at the Week 52 visit. LS means were calculated using a MMRM with baseline fasting blood glucose measurement, stratification factors (country, HbA1c, LDL-C [< 100 mg/dL and ≥ 100 mg/dL], and SU/meglitinide use), treatment, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: 52 weeks
Population: All participants who were randomized, received at least 1 dose of study drug, and had evaluable post-baseline FBG data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 991 | 522
mg/dL | 15.56 (0.38) | 17.08 (0.52)

18. Secondary Outcome: Percentage of Participants With Total and Nocturnal Hypoglycemic Events
Description: A hypoglycemic event is defined by a blood glucose value ≤70 mg/dL (3.9mmol/L). Total hypoglycemic events include documented symptomatic hypoglycemia, asymptomatic hypoglycemia, probable symptomatic hypoglycemia, unspecified hypoglycemia, or severe hypoglycemia. Nocturnal hypoglycemic events refer to any total hypoglycemic event that occurs between bedtime and waking. The percentage of participants was calculated by dividing the number of participants with hypoglycemic or nocturnal hypoglycemic events by the total number of participants analyzed, multiplied by 100.
Time Frame: Baseline to 52 weeks
Population: All participants who were randomized, received at least 1 dose of study drug, and had evaluable hypoglycemia event data.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 1001 | 535
percentage of participants
  Total hypoglycemic events | 77.0 | 79.8
  Nocturnal hypoglycemic events | 48.9 | 59.8

19. Secondary Outcome: Percentage of Participants With HbA1C Equal or Less Than 6.5% and Less Than 7.0 % and Without Nocturnal Hypoglycemia
Description: The percentage of participants with HbA1C ≤ 6.5% or < 7.0% without nocturnal hypoglycemia is presented. Percentage was calculated by dividing the number of participants with the indicated HbA1c values over the total number of participants and multiplying by 100.
Time Frame: Up to 52 weeks
Population: All participants who were randomized, received at least 1 dose of study drug, and had at least 1 post-baseline HbA1c measurement. Missing endpoints were imputed with the LOCF method, using only post-baseline data.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 989 | 523
percentage of participants
  HbA1c ≤ 6.5% | 17.5 | 8.6
  HbA1c < 7.0% | 26.2 | 15.3

20. Secondary Outcome: Percentage of Participants With Equal or Above 2- and 3-fold ULN for Alanine Transaminase/Serum Glutamic Pyruvic Transaminase (ALT/SGPT) and Aspartate Transaminase/Serum Glutamic Oxaloacetic Transaminase (AST/SGOT)
Description: The percentage of participants was calculated by dividing the number of participants equal or above 2- or 3-fold ULN for ALT/SGPT or AST/SGOT by the total number of participants analyzed, multiplied by 100.
Time Frame: Up to 52 weeks
Population: All participants who were randomized, received at least 1 dose of study drug, and had evaluable post-baseline liver enzyme data.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 | Glargine
Number analyzed (Participants) | 990 | 524
percentage of participants
  ≥2-fold ULN for ALT | 6.5 | 4.0
  ≥3-fold ULN for ALT | 1.9 | 0.6
  ≥2-fold ULN for AST | 3.6 | 1.5
  ≥3-fold ULN for AST | 1.0 | 0.4

ADVERSE EVENTS:
Arm/Group | LY2605541 | Glargine
Serious Adverse Events (participants affected / at risk) | 105/1003 | 73/535
Other Adverse Events (participants affected / at risk) | 733/1003 | 390/535
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2605541 (N=1003) | Glargine (N=535)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Angina pectoris (Cardiac disorders) | 3 (3) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 3 (3)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (2) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (3) | 1 (2)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 3 (6) | 5 (8)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 5 (5) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (3)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vestibular ataxia (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (2) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 1 (3) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 5 (5) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Device occlusion (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 4 (5) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (3) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 5 (7) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Gallbladder empyema (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 2 (3)
Pneumonia (Infections and infestations) | 3 (3) | 4 (5)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (4) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (7) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (7) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/453 (1) | 0/227 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/550 (2) | 2/308 (2)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/550 (0) | 1/308 (1)
Prostate cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/550 (0) | 1/308 (1)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Autonomic neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (4) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Complex partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (2) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 3 (4)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1/453 (1) | 0/227 (0)
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 1/453 (1) | 0/227 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vasculitic rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 1 (1)
Glossectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Prostatectomy (Surgical and medical procedures) | 0/550 (0) | 1/308 (1)
Radical neck dissection (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (3) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypoperfusion (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (2) | 0 (0)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2605541 (N=1003) | Glargine (N=535)
Diarrhoea (Gastrointestinal disorders) | 57 (81) | 38 (52)
Nausea (Gastrointestinal disorders) | 37 (51) | 18 (30)
Vomiting (Gastrointestinal disorders) | 35 (49) | 16 (21)
Fatigue (General disorders) | 35 (38) | 14 (15)
Bronchitis (Infections and infestations) | 52 (60) | 24 (26)
Influenza (Infections and infestations) | 59 (68) | 28 (35)
Nasopharyngitis (Infections and infestations) | 141 (196) | 82 (122)
Sinusitis (Infections and infestations) | 38 (51) | 16 (17)
Upper respiratory tract infection (Infections and infestations) | 83 (119) | 33 (48)
Urinary tract infection (Infections and infestations) | 47 (57) | 22 (28)
Weight increased (Investigations) | 26 (28) | 18 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 52 (68) | 20 (47)
Back pain (Musculoskeletal and connective tissue disorders) | 70 (89) | 36 (47)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 42 (50) | 25 (36)
Dizziness (Nervous system disorders) | 32 (36) | 17 (29)
Headache (Nervous system disorders) | 85 (134) | 37 (72)
Cough (Respiratory, thoracic and mediastinal disorders) | 44 (52) | 18 (22)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 34 (40) | 19 (21)
Hypertension (Vascular disorders) | 41 (43) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days